CLINICAL TRIAL: NCT01175772
Title: Maintenance Treatment for Ovarian Carcinoma in Remission by an Antiangiogenic Treatment Strategy With Metronomic/Oral Chemotherapy (Cytophosphan Combined With Low-dose Methotrexate)and COX-2 Inhibition (Celecoxib)
Brief Title: Maintenance Treatment for Ovarian Carcinoma in Remission by an Antiangiogenic Treatment Strategy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to change in the national policy of medications
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0082-09-EMC
Record Dates: First submitted 2010-08-01; First posted 2010-08-05 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Carcinoma
Keywords: Ovary; Carcinoma; Maintenance; Metronomic; Chemotherapy; Time to Progression; overall survival
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma | interventions — Cyclophosphamide; Celecoxib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metronomic Chemoterapy (Experimental): Maintenance Treatment for Ovary Carcinoma by Metronomic Chemotherapy
  Interventions: Drug: Cytophosphan, Celecoxib, Methotrexate

INTERVENTIONS:
Drug: Cytophosphan, Celecoxib, Methotrexate — Metronomic Chemotherapy as maintenance treatment for patients with Ovarian Cancer
  * Cytophosphan tab 50 mg -1x1 per day, continuous
  * Celecoxib tab 200 mg - 1x2 per day, continuous
  * Methotrexate tab 2.5 mg - 1x2 per day, 2 days weekly

SUMMARY:
Preclinical studies showed that metronomic chemotherapy can induce tumor regression secondary to apoptosis of the tumor blood vessels. This effect was increased by combining metronomic chemotherapy with anti-angiogenic drugs. Metronomic chemotherapy has already proved clinical effects too, especially on patients with breast or prostate carcinoma. This study is aimed to test the efficacy of an experimental metronomic chemotherapy regimen in a cohort of patients with ovarian cancer. Patients will receive the proposed regimen as maintenance treatment following response induction by the conventional maximal tolerated dose (MTD) regimen of Carboplatin and Paclitaxel. Our regimen will include Cytophosphan combined with two agents which are expected to act as indirect angiogenic inhibitors: (a) celecoxib, as a selective COX-2 inhibitor and (b) low-dose Methotrexate, as successfully practiced for suppressing the inflammatory manifestations of rheumatoid arthritis. All components of our regimen will be administered orally and continuously for one year based on the hypothesis that its anti-angiogenic properties will be able to suppress the recovery of residual disease, thus extending the time to progression (TTP), and possibly the overall survival as well.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof of papillary-serous ovarian cancer or 1ary peritoneal carcinomatosis.
2. Histological grade III.
3. Original disease in stage III.
4. ECOG performance status: 0-2.
5. Age: 20-80 years.
6. Previous chemotherapy with paclitaxel and carboplatin (only).
7. Previous cyto-reductive surgery.
8. Clinical Complete Response (both physically and by imaging).
9. CA 125 should be either normalized (in at least 50 patients) or while still in decreasing values at monthly measurements.
10. CBC at normal values or with any toxicity at a grade limited to I by NCIC-CTC.
11. Liver and renal functions < 1.5 upper normal limits (UNL) by SMA.
12. The patient's signature on the informed consent.

Exclusion Criteria:

1. Mucinous type ovarian carcinoma.
2. Histological Grade I-II.
3. Current continuous treatment by steroids or by NSAIDs, or by anti-coagulants for "non protocol" reasons.
4. Previous history of active peptic ulcer.
5. Current participation in any other treatment study.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 18 months
  Median time to progression of the cohort will be compared with equivalent measure in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: David Loven, M.D., Study Director — HaEmek Medical Center, Oncology Unit
Locations (1):
- HaEmek Medical Center, Afula, Israel